CLINICAL TRIAL: NCT01555892
Title: Administration of Rapidly Generated EBV-Specific Cytotoxic T-Lymphocytes To Patients With EBV-Positive Lymphoma
Brief Title: Cytotoxic T-Lymphocytes for EBV-positive Lymphoma, GRALE
Acronym: GRALE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other); National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH); Harris County Hospital District (Other Government)
Responsible Party: Principal Investigator, Helen Heslop, Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-29617-GRALE; GRALE (Other: BCM/CAGT); P50CA126752 (NIH)
Record Dates: First submitted 2012-03-13; First posted 2012-03-16 (Estimated); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Hodgkin's Disease; Non-Hodgkin's Lymphoma; Lymphoproliferative Disease; Lymphoma
Keywords: EBV; Hodgkin's Lymphoma; Non-Hodgkin's Lymphoma; Lymphoma Relapse; Autologous or Syngeneic Stem Cell Transplant; T/NK-lymphoproliferative disease; LMP; BARF1; EBNA1
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin; Lymphoproliferative Disorders; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EBV-specific T cells: A (Experimental): Group A: Patients in second or subsequent relapse (or first relapse or with active disease if immunosuppressive chemotherapy contraindicated or multiple relapsed patients in remission who are at a high risk of relapse)** or any patient with primary disease or in first or subsequent remission if immunosuppressive chemotherapy is contraindicated.
  Patients may receive cells with or without lymphodepletion.
  Patients will be treated at Dose Level 3. Each patient will receive 2 injections, 14 days apart, according to the following dosing schedule:
  Day 0: 1 x 10^8 cells/m2
  Day 14: 2 x 10^8 cells/m2
  ** Patients with relapsed or refractory lymphoma that are eligible for a stem cell transplant will not be treated on this study as an alternative to transplant.
  Interventions: Biological: EBV-specific T cells: A
- EBV-specific T cells: B (Experimental): Group B: Patients in remission or with minimal residual disease (MRD) status after autologous or syngeneic SCT.
  Patients may receive cells with or without lymphodepletion.
  Patients will be treated at Dose Level 3. Each patient will receive 2 injections, 14 days apart, according to the following dosing schedule:
  Day 0: 1 x 10^8 cells/m2
  Day 14: 2 x 10^8 cells/m2
  Interventions: Biological: EBV-specific T cells: B

INTERVENTIONS:
Biological: EBV-specific T cells: A — Patients may receive cells with or without lymphodepletion. Dose Level 3: 1 x 10^8 cells/m2 + 2 x 10^8 cells/m2
  Other Names: LMP, BARF1 and EBNA1 specific CTLs
  Arms: EBV-specific T cells: A
Biological: EBV-specific T cells: B — Patients may receive cells with or without lymphodepletion. Dose Level 3: 1 x 10^8 cells/m2 + 2 x 10^8 cells/m2
  Arms: EBV-specific T cells: B

SUMMARY:
Subjects have a type of lymph gland disease called Hodgkin or non-Hodgkin Lymphoma or T/NK-lymphoproliferative disease or severe chronic active Epstein Barr Virus (CAEBV) which has come back, is at risk of coming back, or has not gone away after treatment, including the best treatment we know for these diseases.

Some of these patients show signs of virus that is called Epstein Barr virus (EBV) that causes mononucleosis or glandular fever ("mono" or the "kissing disease") before or at the time of their diagnosis. EBV is found in the cancer cells of up to half the patients with HD and NHL, suggesting that it may play a role in causing Lymphoma. The cancer cells and some immune system cells infected by EBV are able to hide from the body's immune system and escape destruction. We want to see if special white blood cells, called GRALE T cells, that have been trained to kill EBV infected cells can survive in the blood and affect the tumor.

We have used this sort of therapy to treat a different type of cancer called post transplant lymphoma. In this type of cancer the tumor cells have 9 proteins made by EBV on their surface. We grew T cells in the lab that recognized all 9 proteins and were able to successfully prevent and treat post transplant lymphoma. However, in HD and NHL, T/NK-lymphoproliferative disease, and CAEBV, the tumor cells and B cells only express 4 EBV proteins. In a previous study, we made T cells that recognized all 9 proteins and gave them to patients with HD. Some patients had a partial response to this therapy but no patients had a complete response. We then did follow up studies where we made T cells that recognized the 2 EBV proteins seen in patients with lymphoma, T/NK-lymphoproliferative disease and CAEBV. We have treated over 50 people on those studies. About 60% of those patients who had disease at the time they got the cells had responses including some patients with complete responses. This study will expand on those results and we will try and make the T cells in the lab in a simpler faster way. These cells are called GRALE T cells. These GRALE T cells are an investigational product not approved by the FDA.

The purpose of this study is to find the largest safe dose of LMP-specific cytotoxic GRALE T cells created using this new manufacturing technique. We will learn what the side effects are and to see whether this therapy might help patients with HD or NHL or EBV associated T/NK-lymphoproliferative disease or CAEBV.

DETAILED DESCRIPTION:
Subjects (or their syngeneic donor) will give blood for investigators to make EBV-specific (GRALE) T cells in the lab. These cells will be grown and frozen for the subject.

In this study, patients may also receive cyclophosphamide and fludarabine. These two drugs are standard chemotherapy medicines and may be given before the T cells to make space in the blood for the T cells to grow after receiving them. These drugs will be given intravenously daily over three days.

The GRALE T cells will then be thawed and injected into the subject over 1-10 minutes. Initially, two doses of GRALE T cells will be given 2 weeks apart.

If after the 2nd infusion there is a demonstrated partial response or stable disease in the size of the lymphoma on CT or MRI scan as assessed by a radiologist, the subject can receive additional doses of the GRALE T cells if they wish (up to 6 times). Follow up testing will be collected just like after the 1st infusion.

All of the treatments will be given by the Center for Cell and Gene Therapy at Texas Children's Hospital or Houston Methodist Hospital.

We will follow the subjects after the injections. They will either be seen in the clinic or the subject will be contacted by a research nurse yearly for 5 years.

If they receive additional doses of the GRALE T cells as described above, they will be followed until 5 years after the last dose of GRALE T-cells.

ELIGIBILITY:
Inclusion Criteria at time of Procurement

1. Any patient, regardless of age or sex, with EBV-positive Hodgkin's or non-Hodgkin's Lymphoma, (regardless of the histological subtype) or EBV (associated)-T/NK-lymphoproliferative disease or Severe Chronic Active EBV (CAEBV) who may subsequently be eligible for the treatment component
2. EBV positive tumor (can be pending at this time)
3. Weighs at least 12kg
4. Informed consent explained to, understood by and signed by patient/guardian. Patient/guardian given copy of informed consent.

Inclusion Criteria at time of Infusion

1. Any patient, regardless of age or sex, with EBV-positive Hodgkin's or non-Hodgkin's Lymphoma (regardless of histologic subtype), or EBV (associated)-T/NK-lymphoproliferative disease or Severe Chronic Active EBV (CAEBV)* and

   In second or subsequent relapse (or first relapse or with active disease if immunosuppressive chemotherapy contraindicated or multiply relapsed patients in remission who have a high risk of relapse)** OR any patient with primary disease or in first remission if immunosuppressive chemotherapy is contraindicated, e.g. patients who develop Hodgkin disease after solid organ transplantation or if the Lymphoma is a second malignancy e.g. a Richter's transformation of CLL. (Group A)

   OR

   In remission or with minimal residual disease status after autologous or syngeneic SCT. (Group B)
2. EBV positive tumor
3. Patients with bilirubin less than or equal to 3x upper limit of normal, AST less than or equal 5x upper limit of normal, and hemoglobin greater than or equal to 7.0 (may be a transfused value).
4. Patients with a creatinine less than or equal to 2x upper limit of normal for age
5. Pulse oximetry of > 90% on room air
6. Patients should have been off other investigational therapy for 4 weeks prior to entry in this study. PD1/PDL inhibitors will be allowed if medically indicated.
7. Patients with a Karnofsky/Lansky score of greater than or equal to 50
8. Sexually active patients must be willing to utilize one of the more effective birth control methods during the study and for 6 months after the study is concluded. The male partner should use a condom.
9. Informed consent explained to, understood and signed by patient/guardian. Patient/guardian given copy of informed consent.

   * CAEBV is defined as patients with high EBV viral load in plasma or PBMC (> 4000 genomes per ug PBMC DNA) and/or biopsy tissue positive for EBV

     * Patients with relapsed or refractory lymphoma that are eligible for a stem cell transplant will not be treated on this study as an alternative to transplant.

Exclusion Criteria at Time of Procurement

1. Active infection with HIV, HTLV, HBV, HCV (can be pending at this time)

Exclusion Criteria at Time of Infusion

1. Pregnant or lactating
2. Severe intercurrent infection.
3. Current use of systemic corticosteroids > 0.5 mg/kg/day

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2013-01-14 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of toxicity of escalating doses of LMP, BARF1 and EBNA1 T lymphocytes | 8 weeks
  To determine the safety of escalating doses of 2 intravenous injections of autologous or syngeneic rapid LMP, BARF1 and EBNA1 specific T-lymphocytes (VSTs) in patients with EBV-associated Hodgkin's Disease or non-Hodgkin's lymphoma or T/NK-lymphoproliferative disease and CAEBV.

SECONDARY OUTCOMES:
Determine survival and immune function of LMP/BARF1/EBNA1-specific cytotoxic T-lymphocyte lines | 1 year
  To determine the survival and the immune function of LMP/BARF1/EBNA1-specific cytotoxic T-lymphocyte lines
Assess anti-viral and anti-tumor effects of LMP/BARF1/EBNA1-specific EBVST | 1 year
  To assess the anti-viral and anti-tumor effects of LMP/BARF1/EBNA1-specific EBVST

CONTACTS AND LOCATIONS:
Overall Officials: Helen E Heslop, MD, Principal Investigator — Baylor College of Medicine
Locations (3):
- United States (3):
  - Harris Health System (includes ben Taub General Hospital and Smith), Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas

REFERENCES:
- [Derived] Sarathkumara YD, Van Bibber NW, Liu Z, Heslop HE, Rouce RH, Coghill AE, Rooney CM, Proietti C, Doolan DL. Differential antibody response to EBV proteome following EBVST immunotherapy in EBV-associated lymphomas. Blood Adv. 2025 Apr 8;9(7):1658-1669. doi: 10.1182/bloodadvances.2024014937. PMID 39908567
- [Derived] Sharma S, Mehta NU, Sauer T, Rollins LA, Dittmer DP, Rooney CM. Cotargeting EBV lytic as well as latent cycle antigens increases T-cell potency against lymphoma. Blood Adv. 2024 Jul 9;8(13):3360-3371. doi: 10.1182/bloodadvances.2023012183. PMID 38640255